CLINICAL TRIAL: NCT05992701
Title: Effectiveness and Safety of Directional Deep Brain Stimulation for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other); Changhai Hospital, the Second Military Medical University (Unknown); Shenzhen Second People's Hospital (Other); Zhongnan Hospital (Other); West China Hospital (Other); Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua University (Unknown); First Affiliated Hospital of Kunming Medical University (Other); Nanjing Medical University (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-DBS-2101
Record Dates: First submitted 2023-08-01; First posted 2023-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Directional deep brain stimulation (Experimental)
  Interventions: Device: Directional deep brain stimualtion

INTERVENTIONS:
Device: Directional deep brain stimualtion — Directional deep brain stimualtion in the treatment of Parkinson's disease using L305/L306 leads and G107R/G107 implanted pulse generators (Beijing Pins Medical Co.).

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the PINS Deep Brain Stimulation (DBS) system, including the G107R/G107 IPG, L305/L306 directional leads, E204 extensions and related system components.

DETAILED DESCRIPTION:
This is a prospective, open label, non-randomized study. The study will evaluate the clinical outcome and possible adverse effects of the directional DBS treatment. The following data will be collected: therapeutic window, Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III scores, Parkinson's Disease Questionnaire (PDQ-39) summary scores, total electrical energy delivered, the dosage of anti-parkinsonian medications, on time(h/d) without troublesome dyskinesia, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 18 ~ 75;
2. Idiopathic Parkinson's disease;
3. Patient whose symptoms are not adequately controlled by best medical therapy;
4. Hoehn and Yahr stage≥2.5;
5. Patient whose symptoms are improved by at least 30% with levodopa challenge test;
6. Must be an appropriate candidate for the surgical procedures required for bilateral DBS;
7. Is willing and able to comply with all visits and study related procedures;
8. Patient understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

1. Had received lesioning surgical treatment;
2. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception;
3. Any current drug or alcohol abuse;
4. Cognitive impairment (MMSE≦17 for primary school education or MMSE≦24 for middle school education and above);
5. Any significant psychiatric problems, including unrelated clinically significant depression;
6. Any history of craniocerebral injury, tumor, or severe cerebrovascular disease;
7. Severe brain atrophy (confirmed by CT or MRI);
8. A condition requiring or likely to require the use of diathermy;
9. Abnormal blood routine or biochemical test, coagulation dysfunction, serious abnormal liver or kidney function;
10. Uncontrolled high blood pressure, serious heart disease or serious medical or respiratory diseases;
11. Long-term of immunosuppressive or hormone therapy;
12. Other diseases requiring the stimulators;
13. A condition requiring or likely to require the use of MRI;
14. Participated in any other clinical trials within the preceding 3 months;
15. Unwilling or unable to cooperate with the implantation of DBS system;
16. Unwilling or unable to cooperate with postoperative follow-up;
17. Not considered to be applicable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Therapeutic Window | 1 month post the device implanted
  Therapeutic window is the range of stimulation amplitude that produces symptom relief without causing side effects.

SECONDARY OUTCOMES:
Motor Function | 3 months post device-activation
  Change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III score.
Change in PDQ-39 score | 3 months post device-activation
  Using the Parkinson's Disease Questionnaire to acquire a score ranging from 0 to 156 as a summary of all subscores from 39 items. The higher score indicates lower quality of life.
Total Electrical Energy Delivered(TEED) | 3 months post device-activation
  TEED=(Voltage^2×frequency×pulse width)/impedance×1 s
The dosage of anti-parkinsonian medications | 3 months post device-activation
On time(h/d) without troublesome dyskinesia | 3 months post device-activation
Adverse events | 3 months post device-activation

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua University, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Nanjing Brain Hospital Affiliated to Nanjing Medical University, Nanjing
  - Changhai Hospital, the Second Military Medical University, Shanghai
  - Shenzhen Second People's Hospital (the First Affiliated Hospital of Shenzhen University), Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Zhongnan Hospital of Wuhan University, Wuhan

IPD SHARING:
Plan to Share IPD: No